CLINICAL TRIAL: NCT07140666
Title: Analysis of Influence Factors on Osteopenia in Different Treatment of Psoriasis
Status: Completed | Type: Observational
Sponsor: Chongli Yu (Other)
Responsible Party: Sponsor-Investigator, Chongli Yu, PhD Candidate, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2022-196-01-02
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Biologic Therapy; Bone Mineral Density; Osteopenia
MeSH Terms: conditions — Psoriasis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adalimumab: Participants in this group are patients with psoriasis who receive treatment with adalimumab, a TNF-α inhibitor. Adalimumab is a biologic therapy administered by subcutaneous injection and is widely used for moderate-to-severe plaque psoriasis and psoriatic arthritis. This group will be observed to evaluate changes in bone mineral density (BMD) and bone metabolism markers during treatment. Outcomes from this group will be compared with those from other treatment groups to assess the impact of TNF-α blockade on bone health in patients with psoriasis.
- Secukinumab: Participants in this group are patients with psoriasis who receive treatment with secukinumab, an IL-17A inhibitor. Secukinumab is a biologic therapy given by subcutaneous injection, approved for moderate-to-severe plaque psoriasis and psoriatic arthritis. This group will be observed to evaluate changes in bone mineral density (BMD) and bone metabolism markers during treatment. The outcomes will be compared with other treatment groups to assess the influence of IL-17A blockade on bone health in patients with psoriasis.

SUMMARY:
This clinical study aims to evaluate and compare changes in bone mineral density (BMD) and bone metabolism markers in patients with moderate-to-severe psoriasis treated with either Secukinumab or Adalimumab. Psoriasis is a chronic inflammatory disease that may increase the risk of osteoporosis. While biological therapies have shown efficacy in controlling skin lesions, their long-term effects on bone health remain unclear. By assessing lumbar spine and hip BMD and relevant biomarkers over time, this study seeks to clarify the bone-protective or bone-affecting effects of these two commonly used biologic agents. The results may help optimize treatment strategies for psoriatic patients at risk of osteopenia or osteoporosis.

DETAILED DESCRIPTION:
Psoriasis is a chronic, immune-mediated inflammatory skin disease associated with increased systemic inflammation, which may contribute to altered bone metabolism and decreased bone mineral density (BMD). Several studies have reported an elevated risk of osteopenia and osteoporosis in patients with moderate-to-severe psoriasis. The pathophysiological mechanisms may involve pro-inflammatory cytokines, such as TNF-α and IL-17, which influence both skin inflammation and bone remodeling.

Biologic therapies targeting these cytokines have demonstrated significant efficacy in managing psoriasis. However, their long-term impact on bone metabolism and density is still under investigation. Secukinumab, an IL-17A inhibitor, and Adalimumab, a TNF-α inhibitor, are both widely used in clinical practice, but their comparative effects on bone health are unclear.

This prospective, observational, real-world study aims to evaluate the longitudinal changes in BMD (lumbar spine and hip) and bone turnover markers (such as osteocalcin, P1NP, CTX, and iPTH) in psoriasis patients undergoing treatment with Secukinumab or Adalimumab over a follow-up period of XX months. Participants will undergo baseline and follow-up assessments, including dual-energy X-ray absorptiometry (DEXA) and laboratory testing for bone biomarkers.

Key endpoints include:

Changes in BMD at lumbar spine and hip from baseline.

Temporal trends in bone metabolism biomarkers.

Comparison between treatment groups after adjusting for potential confounders (e.g., age, sex, BMI, PASI score, disease duration, inflammatory markers).

Statistical methods such as linear mixed models (LMM), marginal means estimation, and subgroup analysis will be used to evaluate treatment effects. Additional sensitivity analyses including propensity score matching (PSM) and multiple imputation for missing data will be performed to enhance the robustness of findings.

This study is expected to provide clinical evidence on how different biological treatments may influence bone health in psoriatic patients, thus guiding personalized and preventive care strategies for comorbid osteoporosis.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older.
* Clinically confirmed diagnosis of psoriasis (with or without psoriatic arthritis).
* Currently receiving one of the following treatments: TNF-α inhibitor (adalimumab), or IL-17A inhibitor (secukinumab).
* Able and willing to undergo bone mineral density (BMD) assessment using dual-energy X-ray absorptiometry (DXA).
* Signed informed consent provided. Exclusion Criteria
* History of other systemic diseases affecting bone metabolism (e.g., primary hyperparathyroidism, severe chronic kidney disease, Cushing's syndrome).
* Current use of medications known to strongly affect bone metabolism (e.g., long-term corticosteroids, bisphosphonates, denosumab, teriparatide).
* Pregnant or breastfeeding women.
* History of malignancy or other autoimmune diseases requiring systemic immunosuppressive therapy.
* Inability to complete study visits, assessments, or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective cohort study conducted at the Department of Dermatology, First Medical Center of Chinese PLA General Hospital. The study population consists of adult patients diagnosed with psoriasis, with or without psoriatic arthritis, who received clinical care at the dermatology department. Patients were managed with conventional systemic therapies, adalimumab, or secukinumab, and clinical records were reviewed to assess bone mineral density, bone metabolism markers, and related outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Density | Baseline, 6 months, and 12 months
  Bone mineral density will be assessed using dual-energy X-ray absorptiometry (DXA) at the lumbar spine and hip. The primary outcome is the change in BMD compared with baseline, used to evaluate the presence and progression of osteopenia among patients with psoriasis receiving different treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided